CLINICAL TRIAL: NCT07178431
Title: An Open Label Phase I/IIa, Multicenter, Interventional Single-arm Trial of MB-CART 2019.1 in Patients With Refractory Multiple Sclerosis (MS)
Brief Title: MB-CART2019.1 in Refractory Multiple Sclerosis
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Miltenyi Biomedicine GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M-2024-424
Record Dates: First submitted 2025-07-28; First posted 2025-09-17 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Multiple Sclerosis; CAR T Cell Therapy
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MB-CART2019.1 in MS (Experimental): Biological: MB-CART2019.1
  Interventions: Biological: MB-CART2019.1

INTERVENTIONS:
Biological: MB-CART2019.1 — CAR T cell therapy

SUMMARY:
The goal of this trial is to assess the feasibility, safety and preliminary efficacy of MB-CART2019.1 in patients with active refractory primary and secondary progressive MS.

DETAILED DESCRIPTION:
This is a phase l/ll open-label, multicentre, interventional single-arm trial of MB-CART2019.1 in patients with active refractory primary and secondary Multiples Sclerosis.

During the treatment, the patients will undergo a leukapheresis, a lymphodepleting chemotherapy and an administration of the expanded MB-CART2019.1. Phase I is to establish the safety and tolerability of MB-CART2019.1 and to determine a recommended dose for phase IIa (RP2D). During Phase IIa the treatment response after infusion of MB-CART2019.1 as defined by NEDA-3 ("no evident disease activity") will be evaluated. Therefore a BOIN trial design will be used to guide dose escalation and de-escalation decisions in phase I. The second phase will evaluate the efficacy and safety in patients treated with the recommended dose from phase I. The phase II part follows a Simon's 'minimax' two stage design.

ELIGIBILITY:
Inclusion Criteria:

Individuals must meet all of the following criteria to be included in the trial:

1. Have read, understood and signed/dated the informed consent form.
2. Age ≥18 years at the time of screening.
3. Diagnosis of multiple sclerosis fulfilling the 2017 McDonald criteria.
4. Progressive or worsening MS according to 2014 Lublin MS phenotypic criteria
5. Disease activity despite treatment:

   1. Definition for RRMS/SPMS:

      1 or more relapses or an EDSS deterioration in the previous year (1 point or more if EDSS is between 3 and 5.5; 0.5 point or more if EDSS 6-6.5) or MRI activity (presence of at least 2 new/enlarging T2 lesions or T1CE lesions) despite on/previous treatment with an escalation therapy drug (i.e. natalizumab, ofatumumab, ocrelizumab, alemtuzumab or mitoxantrone) for at least 6 months.
   2. Definition for PPMS:

      EDSS deterioration in the previous year (1 point or more if EDSS between 3 and 5.5; 0.5 point or more if EDSS 6-6.5) or MRI activity (presence of at least 2 new/enlarging T2 lesions or T1CE lesions) despite on/previous treatment with ocrelizumab (treatment duration ≥ 6 months).
   3. Evidence of intrathecal IgG production through oligoclonal bands (OCBs) present in the cerebrospinal fluid in PPMS or SPMS.
6. Fully vaccinated against Hepatitis B.
7. Presence of varicella-zoster virus (VZV) antibodies, or completion of at least one dose of varicella zoster glycoprotein E Shingrix vaccine at least 4 weeks prior to treatment.
8. Presence of anti EBV antibodies
9. Organ function / lab parameters as follows

   1. Absolute Neutrophil count > 2000/uL
   2. Platelets > 150,000/uL
   3. Absolute Lymphocyte count > 1000/uL
   4. Serum IgG > 500 mg/dl
   5. Hemoglobin > 9g/dl
10. Adequate renal, hepatic, pulmonary and cardiac function defined as

    1. Creatinine ,< 2mg/dl or creatinine clearance > to 60ml/min
    2. ALT/AST < 3x ULN
    3. Total bilirubin < 1,5 mg/dl, except for subjects with Gilbert syndrome.
    4. Cardiac ejection fraction > 40%, no evidence of significant pericardial effusion (echography) or clinically significant ECG findings
    5. Baseline oxygen saturation > 94% on air room
11. Negative test for Hepatitis B core antibody and Hepatitis C core antibody, CMV, VZ, Herpes simplex virus 1 and 2 ab
12. Negative test for Myelin-Oligodendrocyte-Glycoprotein (MOG) and Aquaporin-4 (AQP-4) autoantibodies
13. Women of childbearing potential (WOCBP) must be able and willing to use at least one highly effective method of contraception from the time of consent until 12 months after the administration of MB-CART2019.1. WOCBP must refrain from donating eggs during the same period. A woman is considered of childbearing potential, i.e., fertile, following menarche and until having been postmenopausal for at least 12 months or unless otherwise permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. For the definition and a list of highly effective methods of contraception, see Appendix 1 Contraception Guidelines.
14. Men whose sexual partners are WOCBP must be able and willing to use at least one highly effective method of contraception (used by themselves or their female partners; see Appendix 1 Contraception Guidelines) from the time of consent until 12 months after the administration of MB-CART2019.1.
15. Willingness and ability to comply with all trial procedures.
16. Adequate vital signs.

Exclusion Criteria:

Patients will be entered into this trial only if they meet none of the following criteria:

1. For relapsing and progressive MS forms: the disability status according to the EDSS scale is larger than 7.0 or the age is larger than 55 years.

   Only applicable for progressive MS (PPMS/SPMS), where the disease duration is longer than 15 years.
2. History of a malignancy unless disease free for ≥5 years with the exception of basal or squamous cell skin cancer
3. Known history of and/or active infection with hepatitis B (hepatitis B surface antigen positive)
4. Known history of infection with hepatitis C virus unless treated and confirmed to be polymerase chain reaction (PCR) negative
5. Any active uncontrolled bacterial, viral or fungal infection
6. A history of and/or active infection with human immunodeficiency virus (HIV)
7. A history of active or latent tuberculosis (TB); TB testing should be performed at screening (Quantiferon test). Confirmed active or latent TB the patient can be re-screened after full completion of anti-tuberculosis treatment (9 months of Isoniazide therapy)
8. History of neuromyelitis optica spectrum disorder (NMOSD) or MOG antibody associated disease.
9. History of CNS or spinal cord tumor, metabolic or infectious causes of myelopathy, genetically inherited progressive CNS disorder, sarcoidosis or non MS-progressive neurological condition affecting the ability to perform the study assessments
10. History of cytopenia consistent with MDS diagnosis
11. History of sickle cell anemia or other hemoglinopathies
12. Primary immune deficiency disease
13. Patients with positive antiphospholipid antibodies, anti-cardiolipin or lupus anticoagulant.
14. History of moderate or worse renal impairment (eGFR < 30 ml/min/1.73 m2)
15. Prevalent inflammatory diseases of the GI tract (e.g. Inflammatory bowel disease, Peptic ulcer) which could result in a higher risk for gastrointestinal perforation.
16. The following cardiac conditions:

    New York Heart Association Stage III or IV congestive heart failure Myocardial infarction or coronary artery bypass graft ≤ 6 months prior to enrollment History of clinically significant ventricular arrhythmia or unexplained syncope, not believed to be vasovagal in nature or due to dehydration
17. History of severe non-ischemic cardiomyopathy Medications:

    Systemic corticosteroids >10 mg within 7 days prior to leukapheresis; T cell targeting drugs (e.g. mycophenolate mofetil, calcineurin inhibitors) within 21 days prior to leukapheresis, Previous CAR T cell therapy, Live vaccines within 30 days prior to leukapheresis, Current Cytotoxic drugs Other MS disease modifying drugs (as stated in 5.8.1.)
18. Hypersensitivity against any drug or its ingredients/impurities that is scheduled or likely to be given during trial participation, e.g. as part of the mandatory preparative lymphodepletion or rescue medication/salvage therapies for treatment related toxicities;
19. Contraindication of trial related procedures as judged by the investigator
20. Pregnant of breast-feeding females; female patients of child-bearing potential not willing to practice a highly effective form of birth control from leukapheresis and for 12 months after dosing the IMP
21. Concurrent participation in another interventional trial
22. Inability to understand the procedures and risks associated with the Trial.
23. Any additional contraindication of trial related procedures as judged by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2030-02-28 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Primary endpoints Phase I | day 28
  * Recommended dose for phase IIa out of 2 dose levels, based on a Bayesian Optimal Interval (BOIN) design, using a target dose limited toxicity (DLT) rate of 30%, with DLT until day 28 after infusion of MB-CART2019.1.
  * Safety and tolerability of MB-CART2019.1 per incidence of adverse event (AE), classified according to CTCAE version 5.0.
  * Evaluation and classification of Cytokine Release Syndrome (CRS) until day 28 after infusion of MB-CART2019.1.
  * Evaluation and classification of Immune Effector cell-associated Neurotoxicity Syndrome (ICANS) until day 28 after infusion of MB-CART2019.1.
Primary endpoints Phase IIa | 48 weeks
  * NEDA-3 ("no evident disease activity") at 48 weeks (fulfilling all of the following):
  * no relapse activity: relapse activity is defined as any new neurologic symptom consistent with MS/not explained otherwise, accompanied by new neurologic signs present for at least 24 hrs.
  * no disease progression in the absence of relapses using a composite endpoint of no 24-week confirmed progression:
  * of ≥1 point/ ≥0.5 point on the EDSS if baseline EDSS ≤5.5/ >5.5 points ;
  * of ≥20% on the timed 25-foot walk test
  * of ≥20%on the 9-hole peg test (NHPT).
  * no MRI activity: MRI activity is defined as:
  * new and/or enlarging T2-hyperintense lesions as detected by MRI (defined as the sum of the individual number of new and/or enlarging T2 lesions at all scheduled at 48 weeks compared to baseline) or
  * new T1-contrast enhancing (CE) lesions as detected by MRI at 12, 24 or 48 weeks compared to baseline.

SECONDARY OUTCOMES:
Secondary endpoints Phase I only (primary in phase IIa) | 48 weeks
  NEDA-3 ("no evident disease activity") at 48 weeks (fulfilling all of the following):
  1. no relapse activity: relapse activity is defined as any new neurologic symptom consistent with MS/not explained otherwise, accompanied by new neurologic signs present for at least 24 hrs
  2. no disease progression in the absence of relapses using a composite endpoint of
     * no 24-week confirmed progression of ≥1 point/ ≥0.5 point on the EDSS if baseline EDSS ≤5.5/ >5.5 points ;
     * no 24-week confirmed progression of ≥20% on the timed 25-foot walk test and
     * no 24-week confirmed progression of ≥20%on the 9-hole peg test (NHPT)
  3. no MRI activity: MRI activity is defined as
     * new and/or enlarging T2-hyperintense lesions as detected by MRI (defined as the sum of the individual number of new and/or enlarging T2 lesions at all scheduled at 48 weeks compared to baseline) or
     * new T1-contrast enhancing (CE) lesions as detected by MRI at 12, 24 or 48 weeks compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Volker Siffrin PD. Dr., Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No